CLINICAL TRIAL: NCT00092651
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, "Factorial" Design Study to Evaluate the Lipid-Altering Efficacy and Safety of Ezetimibe/Simvastatin Combination Tablet in Patients With Primary Hypercholesterolemia
Brief Title: A Study of MK0653A (Ezetimibe (+) Simvastatin) in Patients With Hypercholesterolemia (0653A-038)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653A-038; 2004_048
Record Dates: First submitted 2004-09-23; First posted 2004-09-28 (Estimated); Last update posted 2024-08-23 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
Keywords: Primary hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0653A, ezetimibe (+) simvastatin
Drug: Comparators: simvastatin and ezetimibe

SUMMARY:
The purpose of this study is to evaluate the lipid lowering effects of an investigational drug in patients with hypercholesterolemia (high cholesterol).

DETAILED DESCRIPTION:
The duration of treatment is 4 months.

ELIGIBILITY:
Inclusion Criteria:

* High cholesterol

Exclusion Criteria:

* Patient has a condition which, in the opinion of the investigator, might pose a risk to the patient, interfere with participation in the study, or does not meet the additional criteria as required by the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1398 (Actual)
Dates: Start 2002-09; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Plasma LDL-C | From baseline to study end point, defined in this study as the last available postbaseline LDL-C measurement, after 12 weeks of treatment.

SECONDARY OUTCOMES:
Plasma LDL-C, TG and HDL-C. The proportion of patients achieving LDL-C targets. Tolerability. | From baseline to study end point in TC, TG, HDL-C, ratios of direct LDL-C:HDL-C and TC:HDL-C, non-HDL-C, Apo B, Apo A-I, Apo A-II, Apo E, lipoprotein(a), C[1]reactive protein (CRP), and fibrinogen, after 12 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Bays HE, Ose L, Fraser N, Tribble DL, Quinto K, Reyes R, Johnson-Levonas AO, Sapre A, Donahue SR; Ezetimibe Study Group. A multicenter, randomized, double-blind, placebo-controlled, factorial design study to evaluate the lipid-altering efficacy and safety profile of the ezetimibe/simvastatin tablet compared with ezetimibe and simvastatin monotherapy in patients with primary hypercholesterolemia. Clin Ther. 2004 Nov;26(11):1758-73. doi: 10.1016/j.clinthera.2004.11.016. PMID 15639688
- [Background] Ose L, Shah A, Davies MJ, Rotonda J, Maccubbin D, Tribble D, Veltri E, Mitchel Y. Consistency of lipid-altering effects of ezetimibe/simvastatin across gender, race, age, baseline low density lipoprotein cholesterol levels, and coronary heart disease status: results of a pooled retrospective analysis. Curr Med Res Opin. 2006 May;22(5):823-35. doi: 10.1185/030079906X100131. PMID 16709304
- [Background] Feldman T, Davidson M, Shah A, Maccubbin D, Meehan A, Zakson M, Tribble D, Veltri E, Mitchel Y. Comparison of the lipid-modifying efficacy and safety profiles of ezetimibe coadministered with simvastatin in older versus younger patients with primary hypercholesterolemia: a post Hoc analysis of subpopulations from three pooled clinical trials. Clin Ther. 2006 Jun;28(6):849-59. doi: 10.1016/j.clinthera.2006.06.001. PMID 16860168
- [Background] Feldman T, Ose L, Shah A, Zakson M, Meehan A, Johnson-Levonas AO, Maccubbin D, Tribble DL, Veltri E, Mitchel Y. Efficacy and safety of ezetimibe/simvastatin versus simvastatin monotherapy in hypercholesterolemic patients with metabolic syndrome. Metab Syndr Relat Disord. 2007 Spring;5(1):13-21. doi: 10.1089/met.2006.0033. PMID 18370810
- [Background] Ose L, Reyes R, Johnson-Levonas AO, Sapre A, Tribble DL, Musliner T. Effects of ezetimibe/simvastatin on lipoprotein subfractions in patients with primary hypercholesterolemia: an exploratory analysis of archived samples using two commercially available techniques. Clin Ther. 2007 Nov;29(11):2419-32. doi: 10.1016/j.clinthera.2007.10.004. PMID 18158082
- [Background] Pearson T, Ballantyne C, Sisk C, Shah A, Veltri E, Maccubbin D. Comparison of effects of ezetimibe/simvastatin versus simvastatin versus atorvastatin in reducing C-reactive protein and low-density lipoprotein cholesterol levels. Am J Cardiol. 2007 Jun 15;99(12):1706-1713. doi: 10.1016/j.amjcard.2007.01.062. Epub 2007 May 2. PMID 17560879